CLINICAL TRIAL: NCT06273280
Title: Renal-based Optimization of QUADruple Therapy in Patients With Heart Failure With Reduced Ejection Fraction: a Prospective, Multicentre, International Randomized Study
Brief Title: Renal-based Optimization of QUADruple Therapy in Patients With Heart Failure With Reduced Ejection Fraction.
Acronym: ReQUAD-HF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Collaborators: King Baudouin Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Z-2023025
Record Dates: First submitted 2024-02-14; First posted 2024-02-22 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction
Keywords: heart failure; heart failure with reduced ejection fraction; guideline-directed medical therapy; quadruple therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized-controlled trial. Due to the design, the study is open-label, but the endpoint assessment is blinded.
Who Masked: Outcomes Assessor
Masking Description: Due to the study design, the study is open-label. In order to reduce bias, a study nurse (blinded for allocation arm) will see or call the patient to register the heart failure medication and dose of loop diuretics at three months and optionally 12months (open-label, endpoint-blinded).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Up-titration of GDMT at the discretion of the treating physician.
  Interventions: Procedure: SOC
- Intervention (Experimental): Uptitration of GDMT according to the renal-based approach postulated by the Heart Failure Association of the European Society of Cardiology (HFA-ESC)
  Interventions: Procedure: Protocolized up-titration

INTERVENTIONS:
Procedure: SOC — Physician-guided GDMT up-titration
  Arms: Standard of Care
Procedure: Protocolized up-titration — Renal-based protocolized GDMT up-titration
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to evaluate guideline-directed medical therapy (GDMT) up-titration in patients with heart failure with reduced ejection fraction.The main question it aims to answer is the improvement in prescription rate and dose uptitration of quadruple GDMT in patients with HFrEF, assessed by a weighed composite score.

Participants will be randomized towards control (standard of care, SOC) or intervention group.

Researchers will compare SOC with protocol-based up-titration to see if the protocolized optimization improves prescription rate of GDMT.

ELIGIBILITY:
Inclusion Criteria:

* Left ventricular ejection fraction ≤ 40%, assessed LVEF with imaging within last three months before randomization (TTE/KT/MIBI/MRI)
* NYHA ≥ II

Exclusion Criteria:

* Hemodynamic instability
* Recent acute coronary syndrome (< 1 month before randomisation)
* Already on quadruple heart failure therapy or on triple GDMT in case of eGFR < 30ml/min/1.73m2 or a potassium above 6mmol/L
* eGFR < 20ml/min/1.73², planned for dialysis or already actively treated with chronic dialysis.
* Implantation of a cardiac resynchronization therapy (CRT) within 3 months
* Adult congenital heart disease
* Previous heart transplantation or currently/planned for ventricular assist device
* Women who are pregnant or breastfeeding
* Unable to participate in 3 months follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Weighed composite score of maximal guideline-directed medical therapy | 3 months
  The composite score of maximal guideline-directed medical therapy 3 months after inclusion.(minimum score 0, maximum score 15)

SECONDARY OUTCOMES:
All-cause mortality and heart failure hospitalizations | 3 months
  All-cause mortality and heart failure hospitalization after three months of follow-up
Change in NTproBNP | 3 months
  Change in NT-proBNP over 3 months
Change in renal function | 3 months
  Change in eGFR, calculated with the CKD-EPI formula

OTHER OUTCOMES:
All-cause mortality | 3 months
  All-cause mortality after 3 months
Number of patients with heart failure hospitalizations | 3 months
  Heart failure hospitalizations after 3 months
Change in prescription rate per GDMT class | 3 months
  Uptitration per class of GDMT.
Incidence of predefined safety endpoints | 3 months
  Prespecified safety events (renal function, potassium, hypotension and bradycardia)

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Mullens, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg AV, Genk, Limburg, Belgium